CLINICAL TRIAL: NCT00547768
Title: Comparative Study Evaluating the Effects of Fexofenadine HCI 180 mg With Orange Juice Versus Placebo With Orange Juice in a Skin Wheal and Flare Challenge Model.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M016455A_4144
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fexofenadine HCI

SUMMARY:
Compare the effect of a single dose of fexofenadine HCl 180 mg plus orange juice versus placebo plus orange juice on the change from baseline (pre-dose) in histamine skin flares.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant, non-lactating female subjects; 12-55 years of age; within 15% of normal body weight for their height or had a body mass index (BMI) less than 29.9 kg/m2; positive histamine skin prick tests (or a duplicate histamine skin prick test) of summation flare > 20 mm larger than diluent control, and summation wheal > 6 mm larger than diluent control at the screening Visit 1.

Exclusion Criteria:

* Asthma that required treatment with medication other than an inhaled, short-acting beta agonist
* Signs and symptoms of currently active allergic disease (SAR, perennial allergic rhinitis, episodic allergic rhinitis)
* Upper respiratory tract infection, sinusitis, asthma or flu-like symptoms within 2 weeks prior to Visit 1
* Dermatographism or other skin conditions that might interfere with the interpretation of the skin test results
* Treatment with escalating doses of immunotherapy, oral immunotherapy, or short course (rush) immunotherapy
* Any excessive amounts of alcohol (no more than two drinks/day on average)
* Any excessive use of caffeine (more than six cups of coffee per day or equivalent)
* Any history of chronic alcohol or mood-altering drug abuse
* Any use of tobacco/nicotine products within 90 days of visit 1
* Any disease state or surgery known to affect the gastrointestinal absorption of drugs
* Treatment with an H1-receptor antagonist regularly within the past year before study entry
* Known hypersensitivity to the investigational product or to drugs with similar chemical properties, or to orange juice
* Need to visit a tanning salon during the study
* Need to use artificial tanning products during the study
* Pregnancy
* Breast-feeding
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol (see Section 6.2)
* Treatment with any investigational product in the last 30 days before study entry
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Unlikelihood of complying with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Use of any of the following drugs within the time indicated prior to the first dosing visit (Time prior to Visit 2):
* Systemic or injected corticosteroids (including oral, parenteral, intravenous, rectal)(30 days).
* Nasal or inhaled or ocular corticosteroids (30 days).
* Nasal or inhaled ipratropium bromide (or atropine), inhaled nedocromil, or nasal, inhaled, or ophthalmic sodium cromolyn (14 days)
* Agents with antihistaminic/anticholinergic activity (e.g.antidepressants, antipsychotics)(14 days).
* Leukotriene pathway modifiers (Accolate®, Singulair®, Zyflo®) 10 days Ocular anti-allergy medications including lodoxamide (Alomide®), olopatadine (Patanol®), emedastine difumarate (Emadine®), levocabastine (Livostin®) (10 days).
* Non-steroidal anti-inflammatory ophthalmics including ketorolac (Acular®), flurbiprofen (Ocufen®), suprofen (Profenal®), diclofenac (Voltaren®) (10 days).
* Antihistamines including desloratadine (Clarinex®), loratadine (Claritin®)(10 days).
* Fexofenadine HCl (Allegra®), cetirizine (Zyrtec®), hydroxyzine, azelastine nasal spray (Astelin®), clemastine (7 days)
* Other short-acting antihistamines such as chlorpheniramine or drugs with antihistaminic activity (3 days).
* OTC oral antihistamines, decongestants (includes pseudoephedrine and other decongestants), or antihistamines/decongestant combinations including all cold, cough, and sleep aids (3 days).
* OTC ophthalmic decongestant, antihistamine, or decongestant/ antihistamine combinations (3 days).
* Other anticholinergic agents (3 days).
* Immunotherapy injection (1 day).
* Other drugs were to be permitted if they were not expected to interfere with the ability of the subject to participate in the study.
* Non-steroidal anti-inflammatory agents were not allowed for 2 days prior to each treatment visit day through 24 hours post-dose.
* Medications or agents not specified above that might confound the interpretation of the results were prohibited as follows:
* Caffeine within 6 hours prior to each visit (coffee, tea, cola, including Mountain Dew and Surge).
* Decaffeinated coffee, tea and colas within 6 hours of each visit
* Alcohol within 24 hours prior to each study visit.
* Chocolate within 6 hours prior to each visit.
* Antacids within + 2 hours of investigational product dosing.
* Any waiver of these inclusion and exclusion criteria required approval by the investigator and the sponsor on a case-by-case basis prior to enrolling the subject. Approval had to be documented by both the sponsor and the investigator.
* No subject was to be allowed to enroll in this study more than once.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2002-11; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Size of change in skin flares from baseline measured at pre-specified times post-dose. | 20 min, 40 min, 60 min, and hourly through 12 hours, with an additional 2 time points obtained at Hours 23 and 24.

SECONDARY OUTCOMES:
Size and change in skin wheals from baseline measured at pre-specified time points. | 20 min, 40 min, 60 min, and hourly through 12 hours, with an additional 2 time points.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States